CLINICAL TRIAL: NCT01250730
Title: A Phase 1, Open Label, Dose Escalation, Single Oral Dose Study In Japanese Healthy Male Volunteers To Investigate The Safety, Tolerability And Pharmacokinetics Of PF-02341066
Brief Title: A Study In Japanese Healthy Male Volunteers To Investigate The Safety, Tolerability And Pharmacokinetics Of PF-02341066
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None
Other Study IDs: A8081022
Record Dates: First submitted 2010-11-17; First posted 2010-12-01 (Estimated); Results first posted 2011-11-29 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: PK profile in Japanese healthy male volunteers
MeSH Terms: interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1.0 (Experimental): This study will consist of three cohorts: PF-02341066 150 mg treatment group (n = 6), PF-02341066 250 mg treatment group (n = 6) and PF-02341066 400 mg treatment group (n = 6).
  Interventions: Drug: PF-02341066

INTERVENTIONS:
Drug: PF-02341066 — Cohort 1: a 150 mg single dose of PF-02341066 administered as 1 x 50 mg IRT and 1 x 100 mg IRT.
Drug: PF-02341066 — Cohort 2: a 250 mg single dose of PF-02341066 administered as 1 x 50 mg IRT and 2 x 100 mg IRTs.
Drug: PF-02341066 — Cohort 3: a 400 mg single dose of PF-02341066 administered as 4 x 100 mg IRTs.

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics of single doses of PF-02341066 (150, 250, and 400 mg) in the fasted condition in Japanese healthy male volunteers.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the pharmacokinetics of single doses of PF-02341066 (150, 250, and 400 mg) in the fasted condition in Japanese healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg

Exclusion Criteria:

* Subjects who are smoking,
* Subjects with evidence of disease,
* Subjects with conditions affecting absorption,
* Subjects with treatment with other investigational drug within 30 days,
* Subjects with history of regular alcohol consumption,
* Subjects with use of prescription, nonprescription drugs and dietary supplement within 28 days,
* Subjects with blood donation of approximately 400 mL within 3 months or 200 mL within 1 month prior to dosing

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Hachioji-shi, Tokyo, Japan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081022&StudyName=A%20Study%20In%20Japanese%20Healthy%20Male%20Volunteers%20To%20Investigate%20The%20Safety%2C%20Tolerability%20And%20Pharmacokinetics%20Of%20PF-02341066%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twelve healthy subjects were assigned to open-label crizotinib treatment in either the 150 mg cohort (6 subjects) or 250 mg cohort (6 subjects).
  After the completion of assessment of safety at both 150 mg and 250 mg cohorts, the 400 mg cohort, the highest dose level in this study, was started.
Groups:
- Crizotinib 150 mg: A 150 mg single dose of crizotinib administered as one 50 mg Immediate Release Tablet (IRT) and one 100 mg IRT
- Crizotinib 250 mg: A 250 mg single dose of crizotinib administered as one 50 mg IRT and two 100 mg IRTs
- Crizotinib 400 mg: A 400 mg single dose of crizotinib administered as four 100 mg IRTs.
Period: Overall Study
Arm/Group | Crizotinib 150 mg | Crizotinib 250 mg | Crizotinib 400 mg
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Crizotinib 150 mg | Crizotinib 250 mg | Crizotinib 400 mg | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 18
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero Extrapolated to Infinite Time [AUC(0-inf)] of Crizotinib
Description: AUC(0-inf) of crizotinib is estimated from the crizotinib concentration. It is obtained from AUClast plus (Clast/kel).
  AUClast = area under the plasma concentration-time curve from zero time until the last measurable concentration.
  Clast = the last quantifiable concentration. Kel = terminal phase elimination rate constant.
Time Frame: 0, 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 144 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Crizotinib 150 mg | Crizotinib 250 mg | Crizotinib 400 mg
Number analyzed (Participants) | 6 | 6 | 6
ng*hr/mL | 1423 (471.52) | 3806 (1313.2) | 6569 (2098.3)

2. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of Crizotinib
Description: AUClast of crizotinib is estimated from the crizotinib concentration. It is obtained from Linear/Log trapezoidal method.
Time Frame: 0, 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 144 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Crizotinib 150 mg | Crizotinib 250 mg | Crizotinib 400 mg
Number analyzed (Participants) | 6 | 6 | 6
ng*hr/mL | 1339 (472.66) | 3732 (1312.4) | 6386 (2084.7)

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of Crizotinib
Time Frame: 0, 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 144 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Crizotinib 150 mg | Crizotinib 250 mg | Crizotinib 400 mg
Number analyzed (Participants) | 6 | 6 | 6
ng/mL | 70.54 (25.570) | 155.6 (50.694) | 235.8 (60.988)

4. Primary Outcome: Time to Cmax (Tmax) of Crizotinib
Time Frame: 0, 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 144 hours post-dose
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Crizotinib 150 mg | Crizotinib 250 mg | Crizotinib 400 mg
Number analyzed (Participants) | 6 | 6 | 6
ng/mL | 5.00 [5.00 to 6.00] | 5.00 [4.00 to 6.00] | 5.00 [5.00 to 6.00]

5. Primary Outcome: Terminal Elimination Half-life (t1/2) of Crizotinib
Description: t1/2 of crizotinib is the time measured for the plasma concentration to decrease by one half. It is obtained from a Loge(2)/kel.
  Kel = terminal phase elimination rate constant
Time Frame: 0, 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 144 hours post-dose
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Crizotinib 150 mg | Crizotinib 250 mg | Crizotinib 400 mg
Number analyzed (Participants) | 6 | 6 | 6
hours | 41.08 (6.7683) | 29.90 (3.9945) | 29.13 (3.5753)

6. Primary Outcome: Apparent Oral Clearance (CL/F) of Crizotinib
Description: CL/F of crizotinib is obtained from a Dose per AUCinf.
Time Frame: 0, 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 144 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: liter per hour
Arm/Group | Crizotinib 150 mg | Crizotinib 250 mg | Crizotinib 400 mg
Number analyzed (Participants) | 6 | 6 | 6
liter per hour | 105.4 (33.926) | 65.70 (30.500) | 60.87 (16.936)

7. Primary Outcome: Apparent Volume of Distribution (Vz/F) of Crizotinib
Description: Vz/F of crizotinib is obtained from a Dose / (AUCinf *kel).
  Kel = terminal phase elimination rate constant
Time Frame: 0, 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 144 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: Liter
Arm/Group | Crizotinib 150 mg | Crizotinib 250 mg | Crizotinib 400 mg
Number analyzed (Participants) | 6 | 6 | 6
Liter | 6170 (2843.7) | 2811 (1765.0) | 2545 (958.43)

8. Primary Outcome: Dose Normalized AUC(0-inf) of Crizotinib
Description: Dose normalized (to 150 mg dose) AUC(0-inf) is obtained from AUC(0-inf) / (Dose/150).
Time Frame: 0, 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 144 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Crizotinib 150 mg | Crizotinib 250 mg | Crizotinib 400 mg
Number analyzed (Participants) | 6 | 6 | 6
ng*hr/mL | 1423 (471.52) | 2284 (787.92) | 2463 (786.84)

9. Primary Outcome: Dose Normalized AUClast of Crizotinib
Description: Dose normalized (to 150 mg dose) AUClast is obtained from AUClast / (Dose/150).
Time Frame: 0, 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 144 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Crizotinib 150 mg | Crizotinib 250 mg | Crizotinib 400 mg
Number analyzed (Participants) | 6 | 6 | 6
ng*hr/mL | 1339 (472.66) | 2239 (787.45) | 2395 (781.75)

10. Primary Outcome: Dose Normalized Cmax of Crizotinib
Description: Dose normalized (to 150 mg dose) Cmax is obtained from Cmax / (Dose/150).
Time Frame: 0, 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 144 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Crizotinib 150 mg | Crizotinib 250 mg | Crizotinib 400 mg
Number analyzed (Participants) | 6 | 6 | 6
ng/mL | 70.54 (25.570) | 93.36 (30.416) | 88.41 (22.870)

11. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero Extrapolated to Infinite Time (AUC0-inf) of Plasma Active Metabolite (PF-06260182)
Description: AUC(0-inf) of PF-06260182 is estimated from the PF-06260182 concentration. It is obtained from AUClast plus (Clast/kel).
  AUClast = area under the plasma concentration-time curve from zero time until the last measurable concentration.
  Clast = the last quantifiable concentration. Kel = terminal phase elimination rate constant.
Time Frame: 0, 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 144 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Crizotinib 150 mg | Crizotinib 250 mg | Crizotinib 400 mg
Number analyzed (Participants) | 4 | 6 | 6
ng*hr/mL | 180.8 (99.369) | 535.8 (274.23) | 1046 (549.90)

12. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of Plasma Active Metabolite (PF-06260182)
Description: AUClast of crizotinib is estimated from the crizotinib concentration. It is obtained from Linear/Log trapezoidal method.
Time Frame: 0, 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 144 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Crizotinib 150 mg | Crizotinib 250 mg | Crizotinib 400 mg
Number analyzed (Participants) | 6 | 6 | 6
ng*hr/mL | 188.1 (81.706) | 527.2 (273.68) | 1034 (547.34)

13. Primary Outcome: Maximum Plasma Concentration (Cmax) of Plasma Active Metabolite (PF-06260182)
Time Frame: 0, 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 144 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Crizotinib 150 mg | Crizotinib 250 mg | Crizotinib 400 mg
Number analyzed (Participants) | 6 | 6 | 6
ng/mL | 17.24 (6.2371) | 37.63 (18.372) | 54.94 (14.633)

14. Primary Outcome: Time to Cmax (Tmax) of Plasma Active Metabolite (PF-06260182)
Time Frame: 0, 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 144 hours post-dose
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Crizotinib 150 mg | Crizotinib 250 mg | Crizotinib 400 mg
Number analyzed (Participants) | 6 | 6 | 6
ng/mL | 5.00 [4.00 to 6.00] | 5.00 [4.00 to 6.00] | 6.00 [5.00 to 8.00]

15. Primary Outcome: Metabolite to Parent Ratio AUC(0-inf)
Description: The metabolic ratio (MR) is calculated by first converting the AUC(0-inf) for both crizotinib and metabolite (PF-06260182) from mass units to molar units.
Time Frame: 0, 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 144 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Crizotinib 150 mg | Crizotinib 250 mg | Crizotinib 400 mg
Number analyzed (Participants) | 4 | 6 | 6
ratio | 0.1261 (0.0200) | 0.1365 (0.0272) | 0.1544 (0.0343)

16. Primary Outcome: Metabolite to Parent Ratio AUClast
Description: The metabolic ratio (MR) is calculated by first converting the AUClast for both crizotinib and metabolite (PF-06260182) from mass units to molar units.
Time Frame: 0, 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 144 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Crizotinib 150 mg | Crizotinib 250 mg | Crizotinib 400 mg
Number analyzed (Participants) | 6 | 6 | 6
ratio | 0.1362 (0.0262) | 0.1370 (0.0272) | 0.1571 (0.0347)

17. Primary Outcome: Metabolite to Parent Ratio Cmax
Description: The metabolic ratio (MR) is calculated by first converting the Cmax for both crizotinib and metabolite (PF-06260182) from mass units to molar units.
Time Frame: 0, 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 144 hours post-dose
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Crizotinib 150 mg | Crizotinib 250 mg | Crizotinib 400 mg
Number analyzed (Participants) | 6 | 6 | 6
ratio | 0.2371 (0.0833) | 0.2346 (0.0441) | 0.2260 (0.0429)

ADVERSE EVENTS:
Time Frame: For serious adverse event, up to 28 days after the last administration of the study drugs
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Crizotinib 150 mg | Crizotinib 250 mg | Crizotinib 400 mg
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 0/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crizotinib 150 mg (N=6) | Crizotinib 250 mg (N=6) | Crizotinib 400 mg (N=6)
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.